CLINICAL TRIAL: NCT02332850
Title: A Multi-ARM Phase Ib Study of SAR650984 (Isatuximab, an Anti-CD38 mAb) in Combination With Standard Carfilzomib, and High-dose Weekly Carfilzomib and Dexamethasone for the Treatment of Relapsed or Refractory Multiple Myeloma
Brief Title: Phase Ib Study of SAR650984 in Combination With Carfilzomib for Treatment of Relapsed or Refractory Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Thomas Martin, MD (Other)
Collaborators: Amgen (Industry); Sanofi (Industry)
Responsible Party: Sponsor-Investigator, Thomas Martin, MD, Clinical Professor of Medicine, Division of Hematology/Oncology and Director, Clinical Research, Hematologic Malignancies Program, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 139511; NCI-2015-00712 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2014-12-12; First posted 2015-01-07 (Estimated); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Multiple Myeloma
Keywords: Relapsed; Refractory
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — isatuximab; carfilzomib; Dexamethasone; Calcium Dobesilate; dexamethasone 21-phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (20 mg dexamethasone, isatuximab, carfilzomib) (Experimental): 20 mg dexamethasone IV given on days 1, 8, 15, 22 (pre- SAR650984 and carfilzomib), then dexamethasone 4 IV or PO mg Day 2, 9, 16.
  All patients will receive a fixed dose of Isatuximab (SAR650984) according to their assigned dose cohort. Patients receive isatuximab IV over 4-6 hours on days 1 and 15 of every cycle for the starting cohort, and days 1, 8, 15, and 22 of cycle 1 and days 1 and 15 of subsequent cycles. Carfilzomib IV will be administered over 10 minutes on days 1, 2, 8, 9, 15, and 16 . Treatment repeats every 28 days for 8 courses in the absence of disease progression or unacceptable toxicity. Patients may continue treatment after 8 courses if clinical benefit is present at the investigator's discretion (carfilzomib may be switched to days 1, 2, 15, and 16 after 8 cycles per investigator discretion).
  Interventions: Biological: Isatuximab; Drug: Carfilzomib; Drug: Dexamethasone
- Arm II (40 mg dexamethasone, isatuximab, carfilzomib) (Experimental): 40 mg dexamethasone IV given on Days 1, 8, 15 and 22 (use as premed to isatuximab).
  All patients will receive a fixed dose of Isatuximab (SAR650984) according to the assigned dose. Patients receive isatuximab IV over 4-6 hours on day 1, 3-4 hours on Day 8, 15, and 22 of cycle 1 and then on days 1 and 15 of subsequent cycle (patients may be eligible for rapid siatuximab given over 75 minutes), and carfilzomib IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Isatuximab; Drug: Carfilzomib; Drug: Dexamethasone

INTERVENTIONS:
Biological: Isatuximab — Given IV
  Other Names: SAR 650984
Drug: Carfilzomib — Given IV
  Other Names: Kyprolis; PR-171
Drug: Dexamethasone — Given IV or PO
  Other Names: Orgadrone; Spersadex; Visumetazone

SUMMARY:
This phase Ib trial studies the side effects and best dose of isatuximab when given together with carfilzomib with or without dexamethasone and lenalidomide in treating patients with multiple myeloma that has returned after a period of improvement (relapsed) or has not respond to previous treatment (refractory). Immunotherapy with monoclonal antibodies, such as isatuximab, may induce changes in the body's immune system and may interfere with the ability of tumor cells to grow and spread. Carfilzomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as dexamethasone and lenalidomide, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving isatuximab and carfilzomib with or without dexamethasone and lenalidomide may be a better treatment for patients with multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

ARM 1: To determine the maximum tolerated dose (MTD) of SAR650984 in combination with standard carfilzomib (Arm 1 is complete).

ARM 2: To determine the safety AND efficacy (objective response rate (ORR)) of adding SAR650984 10mg/kg weekly x 4 doses then every other week in combination with weekly carfilzomib (70 mg/m2) and dexamethasone, in patients with relapsed or refractory myeloma. ORR will be defined using the International Myeloma Working Group (IMWG) uniform response criteria.

SECONDARY OBJECTIVES:

ARM 1:

1. To evaluate the safety, including immunogenicity (ARM 1), of SAR650984 in combination with carfilzomib, in patients with relapsed or refractory myeloma after receiving 1+ prior lines of therapy. The severity, frequency and incidence of all toxicities will be assessed.
2. To evaluate the pharmacokinetics (PK) of SAR650984 and carfilzomib when administered in ARM 1 (completed).
3. To assess the relationship between clinical (adverse event and/or tumor response) effects and pharmacologic parameters (PK/PD), and/or biologic (correlative laboratory) results.
4. To estimate the activity (ORR) using the International Myeloma Working Group (IMWG) defined response criteria of SAR650984 plus carfilzomib (ARM 1)
5. To describe progression free survival (PFS), time to disease progression (TTP) and 1-year overall survival (OS) in patients treated with SAR650984 plus standard carfilzomib, and SAR650984 with weekly carfilzomib and dexamethasone.

EXPANSION COHORTS:

ARM 1:

1. To further evaluate safety, PK, PD and to estimate the anti-tumor activity (response rates) using IMWG defined response criteria of study therapy (SAR650984 plus carfilzomib).

ARM 1 and 2:

1. To describe progression-free survival, 1-year OS, and TTP in patients with relapsed or refractory myeloma treated with these combinations.

OUTLINE: This is a dose-escalation study of isatuximab. Patients are randomized to 1 of 2 arms.

ARM I: Patients receive dexamethasone intravenously (IV) on days 1, 8, 15, and 22 of cycle 1, and orally (PO) or IV on days 1 and 15 of subsequent cycles. Patients receive isatuximab IV over 4-6 hours on days 1, 8, 15, and 22 of cycle 1 and days 1 and 15 of subsequent cycles, and carfilzomib IV over 10 minutes on days 1, 2, 8, 9, 15, and 16. Treatment repeats every 28 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity. Patients may continue treatment after 8 cycles if clinical benefit is present at the investigator's discretion (carfilzomib may be switched to days 1, 2, 15, and 16 per investigator discretion).

ARM II: Patients receive dexamethasone IV or PO on days 1, 8, 15, and 22, isatuximab IV over 4-6 hours on 1, 8, 15, and 22 of cycle 1 and days 1 and 15 of subsequent cycles, and carfilzomib IV over 30 minutes on days 1, 8, and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 and 60 days and then every 3 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, age 18 years or older
2. Diagnosis of multiple myeloma (MM) and documentation of treatment

   * ARM 1: Must have prior exposure to an immunomodulatory drug (IMiD) and proteasome inhibitor (PI) and have had 2 prior regimens/lines of therapy; but there is no maximum number of prior regimens, and prior autologous bone marrow transplant is acceptable if > 12 weeks from transplantation; patients may have received prior carfilzomib (sensitive, relapsed and refractory [having progressed while receiving carfilzomib or within 60 days of stopping carfilzomib] are all eligible), but must be > 4 weeks from last dosing of carfilzomib
   * ARM 2: Must have had at least 1 but no more than 3 prior lines of anti-myeloma therapy; may be refractory to lenalidomide but sensitive to carfilzomib; prior exposure to carfilzomib is allowed but may not be refractory to carfilzomib; subjects must be >= 8 weeks from last carfilzomib therapy
   * A line of therapy is defined as a course of therapy that is not interrupted by progressive disease; for example, induction therapy, autologous stem cell transplantation, and maintenance therapy without intervening progressive disease is one line of therapy
3. Confirmed evidence of relapse/disease progression from immediately prior MM therapy or relapsed and refractory to the immediately prior treatment; relapsed and refractory disease is defined as those who are non-responsive (< minimal response) on salvage therapy or experience disease progression within 60 days of last therapy in patients who have achieved an MR or better to previous therapy; relapsed disease is defined as previously treated myeloma that progresses and requires the initiation of salvage therapy but does not meet IMWG criteria for relapsed and refractory
4. Patients may have received prior carfilzomib (sensitive, relapsed and refractory all eligible); response and duration of prior carfilzomib therapy must be known
5. Patients must have measurable disease defined as at least one of the following:

   * Serum M-protein >= 0.5 g/dl (>= 5 g/l)
   * Urine M-protein >= 200 mg/24 hours (h)
   * Serum free light chain (FLC) assay: involved FLC level >= 10 mg/dl (>= 100 mg/l) and an abnormal serum free light chain ratio (< 0.26 or > 1.65)
   * Quantitative immunoglobulin > 500mg/dL for Immunoglobulin A (IgA) or > 500mg/L for Immunoglobulin D (IgD), only for IgA and IgD myeloma (by nephelometry) when the protein electrophoresis under-represents disease burden
   * Biopsy proven plasmacytoma > 1x1 cm (should be measured within 28 days prior to initial investigational agent dosing)
6. Subject has an Eastern Cooperative Oncology Group (ECOG) =< 2 performance status OR Karnofsky >= 60% performance status
7. Females of childbearing potential (FCBP)

   * A female of childbearing potential is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months
   * Females of childbearing potential must have a negative serum beta-human chorionic gonadotropin (beta-hCG) pregnancy test with a sensitivity of at least 50 milli-international units per milliliter(mIU/mL), within 10-14 days of study start (during screening)
   * FCBP must also agree to ongoing pregnancy testing. Pregnancy testing is not required for post-menopausal or surgically sterilized women
   * Females must agree to avoid pregnancy during the study and must agree to use a medically acceptable method of birth control as determined by the study doctor while participating in the study and for at least 5 months after the last dose of study medication
8. Men must agree to use contraception (i.e. a latex condom) during sexual contact with a FCBP even if they have had a successful vasectomy and agree to not donate sperm for 5 months after last study therapy (SAR650984, lenalidomide and carfilzomib).
9. Voluntary written informed consent before performance of any study-related procedure not part of routine medical care with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care
10. Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (in accordance with national and local subject privacy regulations)
11. For patients with platelets > 100,000 cells/ul (100x10^9/L) able to take aspirin daily as prophylactic anticoagulation therapy for ARM 2 (patients intolerant to aspirin may use warfarin, low-molecular-weight heparin or equivalent anti-platelet therapy)
12. Inclusion Clinical Laboratories Criteria. The following laboratory results must be met:

    * Absolute neutrophil count (ANC) > 1,000 cells/dL (1.0 x 10e9/L) (growth factor cannot be used within the previous 7 days)
    * Hemoglobin >= 8.0 g/dl (without transfusion within the previous 7 days)
    * Platelet count > 75,000 cells/dL (75 x 10e9/L)
    * Creatinine clearance >= 30 mL/min (Cockcroft-Gault equation)
    * Serum glutamic oxaloacetic transaminase (SGOT)/aspartate aminotransferase (AST) or serum glutamate pyruvate transaminase (SGPT)/alanine aminotransferase (ALT) < 2.5 x upper limit of normal (ULN)
    * Total bilirubin =< 1.5 x ULN (excluding Gilbert's)
    * Serum calcium (corrected for albumin) level at or below the ULN range (treatment of hypercalcemia is allowed and subject may enroll if hypercalcemia returns to normal with standard treatment) prior to study therapy initiation
    * Left ventricular ejection fraction (LVEF) >= 40% (by echocardiogram or multigated acquisition scan (MUGA) testing)
    * Fasting glucose under control (< 150 mg/dL [8.3 mmol/L])

Exclusion Criteria:

Patients who have met all the inclusion criteria listed above will be screened for the following exclusion criteria:

1. Diagnosed or treated for another malignancy within 3 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, low-risk prostate cancer after curative therapy or complete resection of other advanced malignancy with the expectation that the patient has received curative therapy
2. Patient has received other investigational drugs with 21 days before enrollment (or must be > than four half-lives of the experimental agent); no prior SAR650984 anti-CD38 antibody therapy allowed
3. History of significant cardiovascular disease unless the disease is well-controlled or history of myocardial infarction in the past 6 months; significant cardiac diseases includes second/third degree heart block; significant conduction abnormalities, significant ischemic heart disease; poorly controlled hypertension; congestive heart failure of New York Heart Association (NYHA) class II or worse (slight limitation of physical activity; comfortable at rest, but ordinary physical activity results in fatigue, palpitation, or dyspnea) and inability to tolerate intravenous hydration necessary for study therapy administration
4. Prior autologous or allogeneic peripheral stem cell transplant within 12 weeks of the first dose of study treatment
5. Daily requirement for corticosteroids (> 10 mg prednisone once daily (QD) or equivalent)
6. Patients with evidence of significant mucosal or internal bleeding
7. Prior radiation therapy or chemotherapy within 2 weeks or major surgical procedure within 4 weeks of the first dose of study treatment
8. Known active infection requiring parenteral or oral anti-infective treatment, once a patient has completed antibiotics and symptoms of infection have resolved to < grade 2, they are then considered eligible from an infection standpoint
9. Serious psychiatric illness, active alcoholism, or drug addiction that may hinder or confuse follow-up evaluation
10. Any medical conditions that, in the Investigator's opinion, would impose excessive risk to the patient; examples of such conditions include any pre-existing kidney disease (acute or chronic, unless renal insufficiency is felt to be secondary to MM), hypertension, active seizure disorder or pulmonary diseases that would impose excessive risk to the patient
11. Patient has hypersensitivity to boron, mannitol sucrose, histidine (as base and hydrochloride salt) and polysorbate 80 or any of the components of study therapy including required prophylactic medications
12. Known human immunodeficiency virus (HIV) seropositivity or active hepatitis B or C viral infection
13. Neuropathy >= grade 3 or painful neuropathy >= grade 2 (National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] version [v]4.03)
14. Gastro-intestinal abnormalities, including bowel obstruction, inability to take oral medication, requirement for intravenous (IV) alimentation, active peptic ulcer or prior surgical procedures or bowel resection affecting absorption

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2015-01-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
ARM I: Incidence of Dose-Limiting Toxicities (DLT) | Up to 60 days of the last dose of study drug
  Treatment-related Adverse events resulting in a DLT will be summarized by maximum toxicity grade for each dose level of isatuximab.
ARM I: Maximum tolerated dose (MTD) of isatuximab | At the end of Cycle 1 (each cycle is 28 days)
  The MTD is defined as the dose level below the lowest dose that induces dose- limiting toxicity in at least one-third of patients Adverse events will be summarized by maximum toxicity grade and by dose level for each ARM of the trial using NCI CTCAE v4.03
ARM II: Overall Response Rate (ORR) | Up to 60 days of the last dose of study drug
  Overall response rate (ORR) as define by the International Myeloma Working Group (IMWG) uniform response criteria of patients obtaining Stringent Complete Remission (sCR), Complete Remission (CR), Very Good Partial Remission (VGPR), Partial Remission (PR), or Minimal Remission (MR)

SECONDARY OUTCOMES:
ARM I: Pharmacokinetic (PK) profile of isatuximab | Baseline, 2 hours mid-infusion, 4, 7, and 11 hours after end of infusion on day 1, days 2, 3, 8, and 15 of course 1, and 0 and 4 hours after end of infusion on day 1 of courses 2-8 (and 0 hours on day 15 of course 2 only)
  Individual plasma concentrations and PK parameters of SAR650984 will be tabulated with standard descriptive statistics. Pharmacokinetic analyses will be carried out in the Pharmacokinetics, Dynamics and Metabolism Department at Sanofi for SAR650984 and carfilzomib.
ARM I: Overall Response Rate (ORR) | Up to 60 days of the last dose of study drug
  Overall response rate; defined as sCR+CR+VGPR + PR utilizing IMWG Uniform Response Criteria
ARM I: Clinical benefit response (CBR) | Up to 60 days of the last dose of study drug
  defined as CR + VGPR + PR + minor response (MR), utilizing International Myeloma Working Group (IMWG) Uniform Response Criteria
ARM I: Incidence of isatuximab-specific antidrug antibodies (ADA) | Up to 1 year
  Analysis of Incidence of isatuximab-specific antidrug antibodies (ADA) to be performed by Sanofi-Oncology.
ARM I: Percentage of bone marrow cells expressing cell surface determinant, CD38 and receptor density | Up to 30 days of the last dose of study drug
  The overall percentage of bone marrow cells expressing cell surface determinant, CD38 and receptor density will be reported.
Overall survival (OS) | assessed at 1, 2, and 3 years from start of treatment
  Duration of time from start of treatment to death on study from any cause,
Progression Free Survival (PFS) | from start of treatment up to 1 year
  Duration of time from start of treatment to the first occurrence of disease progression or death on study from any cause, whichever occurs earlier,
Time To Progression (TTP) | from start of treatment up to 1 year
  Defined as the duration from start of treatment until the first occurrence of disease progression with deaths from causes other than disease progression, censored
Duration of Response (DOR) | up to 60 days of the last dose of study drug
  The duration of overall response is defined as the time period when criteria are met for MR or better (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented. The duration of CR is defined as the time when criteria are first met for CR until the first date that IMWG relapse is objectively documented
Changes in pharmacodynamics variables as they relate to dose, response, and toxicity of carfilzomib in combination with isatuximab | Baseline to up to 30 days of the last dose of study drug
  Changes from baseline in pharmacodynamic markers and proliferation markers, will be evaluated and summarized for each dose cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Martin, MD, Principal Investigator — University of California, San Francisco
Locations (6):
- United States (5):
  - University of California, San Francisco, San Francisco, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Sarah Cannon Cancer Center, Nashville, Tennessee
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No